CLINICAL TRIAL: NCT06135389
Title: Population Pharmacokinetics of Paracetamol in Overweight and Obese Children
Acronym: PARAENFO
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 201129; 2022-A01743-40 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2023-07-12; First posted 2023-11-18 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Overweight; Obesity
Keywords: Obesity; Overweight; population pharmacokinetics; paediatrics
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- blood sampling scheme1: 3 strata of 10 children and adolescents - normal weight, overweight and obese Titration of paracetamol (acetaminophen) - scheme 1
  Interventions: Biological: Titration of paracetamol and its metabolites - scheme1
- blood sampling scheme2: 3 strata of 10 children and adolescents - normal weight, overweight and obese Titration of paracetamol (acetaminophen) - scheme 2
  Interventions: Biological: Titration of paracetamol and its metabolites - scheme 2

INTERVENTIONS:
Biological: Titration of paracetamol and its metabolites - scheme1 — 15 to 20 minutes and 1 to 2 hours after first perfusion and before second perfusion/administration of paracetamol
  Groups: blood sampling scheme1
Biological: Titration of paracetamol and its metabolites - scheme 2 — 30 to 40' after first perfusion and before second perfusion/administration of paracetamol (residual concentration)
  Groups: blood sampling scheme2

SUMMARY:
The main objective of the study is to define population pharmacokinetic parameters and variability factors for paracetamol and its metabolites in overweight and obese children compared to children with normal weight for age and sex.

DETAILED DESCRIPTION:
This study will determine the pharmacokinetic parameters of paracetamol and its metabolites in overweight and obese children compared to children with normal weight for age and sex. The results will enable establishing dosage recommendations for paracetamol in overweight and/or obese children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6 to 17 inclusive with normal weight for age and gender (body mass index [BMI]<25kg/m2 adult equivalent at 18 years [IOTF 25]), overweight (body mass index [BMI]≥ 25kg/m2 adult equivalent at age 18 [IOTF 25] and obese (BMI ≥ 30kg/m2 adult equivalent at age 18 [IOTF 30]) for age and sex
* Surgical procedure requiring treatment with paracetamol intravenously as an analgesic
* No opposition by the holder(s) of parental authority

Exclusion Criteria:

* History of chronic anaemia (≤ 5g/100ml)
* History of hepatocellular insufficiency (ASAT, ALAT ≥ 3N)
* History of renal impairment (<60mL/min*1.73m2)
* History of Gilbert's disease
* History of Type 2 diabetes
* Major motor or neurological disability
* Intake of paracetamol within 24 hours before study inclusion (injection of paracetamol IV or oral intake)
* Patients treated with medicinal products known to affect CYP2E1 or UGT (UDP glucuronosyltransferase): isoniazid, antiepileptic drugs (carbamazepine, phenytoin or phenobarbital), antiretroviral and tyrosine kinase inhibitors

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Non-obese, overweight and obese children aged 6 to 17 scheduled for surgery requiring intravenous (IV) paracetamol injection intraoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of paracetamol and its metabolites: glucuronide, sulfoconjugate, cysteine- and mercapturate-conjugates after a single intravenous perfusion of paracetamol | 2 hours
  The overall concentrations (parent drug and metabolites) have the same unit

SECONDARY OUTCOMES:
Aspartate aminotransferase (ASAT) (UI/L) | 24 hours
  Liver function tests
Alanine aminotransferase (ALAT) (UI/L) | 24 hours
  Liver function tests
Alkaline Phosphatase PALK (UI/L) | 24 hours
  Liver function tests
Bilirubin (μmol/L) | 24hours
  Liver function tests
Gamma-Glutamyl transpeptidase (UI/L) | 24 hours
  Liver function tests

CONTACTS AND LOCATIONS:
Overall Officials: Sihem BENABOUD, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré University Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No